CLINICAL TRIAL: NCT04125199
Title: Effects of Decohexaenoic Acid Supplementation on Markers of Inflammatory Muscle Damage Induced by Eccentric Exercise in Endurance Athletes
Brief Title: Effects of Decohexaenoic Acid Supplementation on Markers of Inflammatory Muscle Damage
Acronym: (EDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCAMCFE-0009
Record Dates: First submitted 2019-09-05; First posted 2019-10-14 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Sport

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Dietary Supplement: supplement consumption
- control group (Placebo Comparator)
  Interventions: Dietary Supplement: supplement consumption

INTERVENTIONS:
Dietary Supplement: supplement consumption — Composition of the Experimental Product: Concentrated oil of Tridocosahexaenoin-AOX® * (350 mg per capsule), α-tocopherol and coating agent (gelatin). Each capsule is 700 mg, of which 500 mg is oil.
  Placebo composition: Olive oil (each capsule is 700 mg).
  Number of capsules: 6 per day, for any of the two products. The dose taken daily is 2.1 g / day for DHA.
  Supplementation Period: Each group completed two 10-week consumption periods for each of the products, with an intermediate washing period of 4 weeks (28 days).

SUMMARY:
Randomized, placebo-controlled, double-blind, placebo-controlled clinical trial consisting of 15 triathletes in which it is intended to observe less inflammatory damage at the muscular level after performing eccentric exercises.

ELIGIBILITY:
Inclusion Criteria:

* Male sex.
* Age: between 18 and 45 years.
* BMI ≤ 35 Kg / m2.
* Volunteers capable of understanding the clinical study, competent to grant written informed consent and willing to comply with the study procedures and requirements.
* Subjects who do not suffer from chronic diseases.
* Non-smoking subjects or less than 10 cigarettes a day.
* Subjects who have not consumed any type of NSAID within 48 hours prior to the study or during its development.
* Subjects without a history of administration of corticosteroids the previous month or during the study.
* Subjects without allergy to any of the products under investigation.
* Patients who have not modified their habits in the performance of physical activity during the study (injuries, injuries ...).
* Patients who have not modified their dietary habits during the previous month or intend to do so during the study.

Exclusion Criteria:

* Subjects who do not consume medication or nutritional supplements with antioxidant and / or anti-inflammatory properties.
* Subjects who do not consume diets with abundant antioxidant and / or anti-inflammatory products.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | It was measured before and after consumption of the supplement. In each of the times it was measured four times. Before performing the eccentric exercises, just after, at 24 and 48 hours later.
  Changes in the inflammatory marker: C-reactive protein (ml / dl). It is measured in venous blood by blood extraction.

SECONDARY OUTCOMES:
muscle damage | It was measured before and after consumption of the supplement. In each of the times it was measured four times. Before performing the eccentric exercises, just after, at 24 and 48 hours later.
  Changes in markers of muscle damage will be measured by serum lactate dehydrogenase (IU / L)
connective tissue injury | It was measured before and after consumption of the supplement. In each of the times it was measured four times. Before performing the eccentric exercises, just after, at 24 and 48 hours later.
  changes in markers of connective tissue injury: serum collagenase. They will be measured by blood extraction.
Hematological variables: LEUCOCITS AND PLATES | It was measured before and after supplement consumption. In each of the times it was measured four times. 1: before performing the eccentric exercises, 2: just after, 3: at 24 hours after and 4: 48 hours later.
  changes in the hematological profile. The samples are analyzed by the laboratory analyzer: BA 400 BioSystems
Biochemical variables | It was measured before and after consumption of the supplement. In each of the times it was measured four times. Before performing the eccentric exercises, just after, at 24 and 48 hours later.
  changes in lipid profile: : basal glycemia(mg/dl), lipid profile: total cholesterol (mg / dl), high density lipoprotein (mg / dl), low density lipoprotein (mg / dl), triglycerides (mg / dl), atherogenic index.
Variable for the evaluation of fatigue: Subjective perception test of Borg's effort | at the end of the stress test with the multipower. It was measured three times. 1: at the end of the test, 2: at 24 hours, 3: at 48 hours.
  change in the perception of fatigue
Perception of pain through the analog visual scale. | at the end of the stress test with the multipower. It was measured three times. 1: at the end of the test, 2: at 24 hours, 3: at 48 hours.
  changes in the perception of muscle pain. Muscle pain will be measured from 0 (no pain), to 10 (unbearable pain).
Isokinetic variables | Twice. One, before the consumption of the product under study and another after the consumption of the product. It was measured after 10 weeks.
  changes in isokinetic variables: Peak torque, peak torque or force moment in extension and flexion in the different muscles involved and at the different measurement moments .It is measured in volts.
Anthropometric variables | Two measurements. One, before the consumption of the product under study and another at 8 weeks of product consumption.
  Weight (Kg), size (cm), BMI kg / m2. Perimeters (measured in cm): (waist, hip, waist / hip index, relaxed biceps, contracted biceps, medial thigh, twin or calf).Folds (mm) (tricipítal, subscapular, suprailiac anterior or supraspinal, abdominal, quadricipital or thigh, leg or calf medial, bicipital, iliocrestal).
  Diameters (cm) (radiocubital or wrist biestiloid, humeral or elbow bicpicondiolo, femoral or knee bicondiol).
Impedancemetric variables | Two measurements. One, before the consumption of the product under study and another at 8 weeks of product consumption.
  fat mass, total water, lean mass (measured in%), muscle mass, bone mass (kg), basal metabolism (KJ).
liver safety variables | It was measured before and after consumption of the supplement. In each of the times it was measured four times. Before performing the eccentric exercises, just after, at 24 and 48 hours later. One year
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No